CLINICAL TRIAL: NCT00650910
Title: An Open-Label, Two-Part, Single Sequence Study to Examine the Effects of Lapatinib on the Pharmacokinetics of Orally Administered Digoxin in Subjects With Metastatic ErbB2 Positive Breast Cancer
Brief Title: Study To Examine The Effects Of Lapatinib On The Pharmacokinetics Of Digoxin In Subjects w/ ErbB2 Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF110557
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms, Breast
Keywords: lapatinib; Metastatic ErbB2 positive breast cancer; digoxin
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lapatinib + digoxin (Experimental): All subjects received 0.5mg digoxin on Days 1 and 9 with daily dosing of 1500mg oral lapatinib starting on Day 2 and continuing through Day 9. Subjects could continue past Day 9 on daily oral lapatinib until Week 10 when they could transfer into a rollover study (EGF19060 or EGF111767).
  Interventions: Drug: lapatinib; Drug: Digoxin

INTERVENTIONS:
Drug: lapatinib — 1500 mg oral lapatinib starting Day 2 continuing through Day 9. Part 2 subjects received 1500mg daily through week 10.
Drug: Digoxin — 0.5mg on Days 1 and 9
  Other Names: lapatinib

SUMMARY:
This is a two part study looking at the effect of lapatinib on concentrations of digoxin in the blood when both drugs are dosed together in Part 1; and looking at the safety and antitumor effect of lapatinib when used together with possible additional anticancer therapy as chosen at the doctor's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, histologically confirmed breast cancer that overexpresses ErbB2 (3+ by IHC, FISH, or CISH positive).
* Is at least 18 years of age and not greater than 65 years of age.
* Is male or female.
* A female is eligible to enter and participate in the study if she is of:

  - Non-childbearing potential (i.e. physiologically incapable of becoming pregnant), including any female who:
* Has had a hysterectomy
* Has had a bilateral oophorectomy (ovariectomy)
* Has had a bilateral tubal ligation, or
* Is post-menopausal (a demonstration of total cessation of menses for ≥ 1 year) or

  - Childbearing potential, has a negative serum pregnancy test at Screening and agrees to one of the following:
* Double-barrier contraception (condom with spermicidal jelly, foam, suppository, or film; diaphragm with spermicide; or male condom and diaphragm).
* Complete abstinence from sexual intercourse from two weeks prior to administration of the study drug, throughout the active study treatment period, and through the Week 10 Visit.
* Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
* Is able to swallow and retain oral medication.
* ECOG performance status 0 to 2.
* Provided written informed consent.
* Adequate bone marrow function.
* Clinical lab results with ranges as stated per protocol.
* Potassium and magnesium within the normal range of institutional values. [Serum potassium or magnesium values that fall outside the normal range may be repeated once at the discretion of the investigator, provided they are considered to be clinically insignificant.]
* Has a left ventricular ejection fraction (LVEF) within the normal institutional range based on ECHO or MUGA.
* Life expectancy of at least 12 weeks
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Is pregnant or lactating.
* Has malabsorption syndrome, a disease affecting gastrointestinal function, or resection of the stomach or small bowel.
* Has evidence of symptomatic or uncontrolled brain metastases or leptomeningeal disease. Subjects with brain metastases treated by surgery and/or radiotherapy are eligible if neurologically stable and do not require steroids or anticonvulsants.
* Is considered medically unfit for the study by the investigator as a result of the medical interview, physical exam, or screening investigations.
* Has CTCAE Grade 2 or greater hypercalcemia as per protocol.
* Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to digoxin or drugs chemically related to the investigational product such as gefitinib [Iressa] and erlotinib [Tarceva].
* Has received treatment with any investigational drug in the previous four weeks.
* Has received chemotherapy, immunotherapy, biologic therapy or hormonal therapy for the treatment of cancer within the past 14 days, with the exception of mitomycin C which is restricted for the past six weeks.
* Is currently receiving amiodarone or has received amiodarone in the six months prior to screening.
* Is receiving any prohibited medication within the timeframe indicated on the prohibited medication list as per protocol.
* Has physiological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Subjects with certain disorders involving heart failure associated with preserved left ventricular ejection fraction such as restrictive cardiomyopathy, constrictive pericarditis, amyloid heart disease, acute cor pulmonale, idiopathic hypertrophic subaortic stenosis, or any other cardiac condition that would preclude the administration of digoxin.
* Has a clinically significant electrocardiogram (ECG) abnormality, including but not limited to sinus node disease, pre-existing incomplete AV block, and Wolff Parkinson-White Syndrome.
* Has inadequate venous access for protocol-related blood draws.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-04-23 (Actual); Primary Completion 2009-07-10 (Actual); Study Completion 2009-07-10 (Actual)

PRIMARY OUTCOMES:
To characterize the effect of repeat oral dose lapatinib treatment on the pharmacokinetics of a single oral dose of digoxin in adult subjects with metastatic ErbB2 positive breast cancer. | 10 days

SECONDARY OUTCOMES:
Safety and tolerability assessments including evaluation of adverse events (AEs) and changes in laboratory values, and vital signs. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Albuquerque, New Mexico, United States
- GSK Investigational Site, Edmonton, Alberta, Canada
- South Korea (2):
  - GSK Investigational Site, Seodaemun-gu, Seoul
  - GSK Investigational Site, Seoul

REFERENCES:
- See also: Results for study EGF110557 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/EGF110557?search=study&search_terms=110557#rs